CLINICAL TRIAL: NCT05527652
Title: Self-Supporting Nasopharyngeal Airway (ssNPA) Treating Upper Airway Obstruction in Hypotonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Zopf, Adjunct Associate Professor of Otolaryngology-Head and Neck Surgery, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00220966; 1R61HL151952 (NIH)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obstructive Sleep Apnea; Hypertonia, Muscle; Nasal Airway Obstruction; Tolerance; Trisomy 21; Down Syndrome
Keywords: Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Hypertonia, Muscle; Apnea; Respiration Disorders; Respiratory Tract Diseases; Sleep Disorders, Intrinsic; Dyssomnias; Sleep Wake Disorders; Nervous System Diseases; Neuromuscular Manifestations; Neurologic Manifestations
MeSH Terms: conditions — Sleep Apnea, Obstructive; Muscle Hypertonia; Nasal Obstruction; Down Syndrome; Sleep Apnea Syndromes; Apnea; Respiration Disorders; Respiratory Tract Diseases; Sleep Disorders, Intrinsic; Dyssomnias; Sleep Wake Disorders; Nervous System Diseases; Neuromuscular Manifestations; Neurologic Manifestations

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 to receive (1) immediate therapy with the ssNPA device or (2) a waitlist control group who will receive standard of care (SoC) for the first 8 weeks and then be offered the ssNPA at week 8 for the rest of the study period (till week 16).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Aggregate and stratified outcomes will be revealed only to the unblinded statisticians with a firewall related to outcomes between statistician and investigators. Dr. Zopf will be blinded to all aggregate/stratified outcomes and Dr. O'Brien will be blinded to polysomnography and quality of life outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Self-Supporting Nasopharyngeal Airway (ssNPA) (Experimental)
  Interventions: Device: Self-Supporting Nasopharyngeal Airway (ssNPA)
- Standard of Care (No Intervention): Waitlist control group: While waiting, participants will continue to receive the treatment they would have had before which will likely include being placed on the waiting list for positive airway pressure (PAP). After a period of being on the waitlist (8 weeks) there is an option to cross-over to the device arm.

INTERVENTIONS:
Device: Self-Supporting Nasopharyngeal Airway (ssNPA) — The ssNPA device is made of a single piece of flexible, medical-grade silicone. It is inserted through one nostril and extends to the anatomic position bypassing the upper airway obstruction above the epiglottis.
  Arms: Self-Supporting Nasopharyngeal Airway (ssNPA)

SUMMARY:
The researchers are investigating if the Self-Supporting Nasopharyngeal Airway (ssNPA) device can be used in the treatment of obstructive sleep apnea in children with Hypotonic Upper Airway Obstruction (HUAO).

ELIGIBILITY:
Inclusion Criteria:

* Children with Hypotonic Upper Airway Obstruction (HUAO): This includes those who newly diagnosed with obstructive sleep apnea (OSA). These children will undergo overnight polysomnography to determine the presence of OSA (apnea-hypopnea index [AHI]>10 or AHI>5 with nocturnal hypoxemia defined as oxygen saturation by pulse oximetry [SpO2] nadir <=75%).
* All subjects require the presence of at least one symptom of OSA (such as snoring 3 or more nights per week, daytime sleepiness, or hyperactive/inattentive behaviors)
* Post adenotonsillectomy or those with contraindications to tonsillectomy.
* Tonsil size 2+ or smaller.
* Parent/caregivers willing and able to provide informed consent and child willing and able to provide assent, where appropriate.

Exclusion Criteria:

* AHI ≤10 on polysomnogram (PSG) without hypoxemia or AHI<5 with hypoxemia.
* Any medical reason why Self-Supporting Nasopharyngeal Airway (ssNPA) therapy may not be suitable
* Active Coronavirus (COVID) 19 infections
* End-tidal carbon dioxide (ETCO2) or Transcutaneous carbon dioxide (TCO2) values >60 mmHg for >10% of sleep time on PSG
* Psychiatric, medical, or social factors likely to invalidate assessments, make adherence with ssNPA highly unlikely or make local follow-up at 8 weeks unfeasible. Some psychiatric conditions may be provoked or exacerbated by OSA, and those most commonly implicated - Attention Deficit/Hyperactivity Disorder, Conduct Disorder, and Oppositional Defiant Disorder - will not be exclusions. However, more pervasive conditions such as severe autism will be excluded.
* Presence of supraglottic airway collapse or more distal airway stenosis or collapse (for example glottic, subglottic stenosis, or concern for distal airway stenosis or malacia)
* Moderate/severe tracheobronchomalacia
* Need for anticoagulative therapy
* Bleeding disorder
* Restrictive thoracic disorders

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | Up to 16 weeks
  Measured during the polysomnogram
Self-Supporting Nasopharyngeal Airway (ssNPA) tolerance | Up to 16 weeks
  Measured by self report. Likert scale 0-5 (higher score is better)

SECONDARY OUTCOMES:
Sleep quality | Up to 16 weeks
  Higher score in parent report of sleep quality on scale 0-5 (higher score is better)
Snoring frequency | Up to 16 weeks
  As reported by participant/care taker in survey given daily. Snoring frequency is rated on a Likert scale 1-5 where 5 indicates snoring more frequently.
Daytime sleepiness | Up to 16 weeks
  Measured using the children's Epworth Sleepiness Scale - The Epworth Sleepiness Scale is a self-administered form with eight items investigating sleep propensity in different real-life situations during the preceding months. Each item can received 0-3 points, thus the final score ranges from 0 (best score) to 24 (worse score).
Quality of life as indicated by the dimensions of the PedsQL (pediatric quality of life) instrument. | Up to 16 weeks
  There are several dimensions of the PedsQL: Physical Functioning, Emotional Functioning, Social Functioning and School Functioning. Each domain will be scored on a scale of 0 (never have problems) to 4 (almost always have problems) and transformed on a scale of 0-100 by reverse scoring (0=100, 1=75, 2=50, 3=25, 4=0). Psychosocial Health Summary Score is the sum of the items over the number of items answered in the Emotional, Social, and School Functioning scales. Physical Health Summary Score is the Physical Functioning Scale Score. The total quality of life score is the sum of all the items over the number of items answered on all scales.

CONTACTS AND LOCATIONS:
Overall Officials: David A Zopf, MD, Principal Investigator — The University of Wisconsin; Louise M O'Brien, PhD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No